CLINICAL TRIAL: NCT05230745
Title: ContraBand™ Safety & Feasibility Study for Treatment of Heart Failure
Brief Title: ContraBand™: Safety & Feasibility Study (RM-20-01)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restore Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-20-01
Record Dates: First submitted 2022-01-05; First posted 2022-02-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure, Left Sided
Keywords: pulmonary artery banding
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ContraBand implants (Experimental): Percutaneous implantation of the ContraBand devices by right heart catheterization
  Interventions: Device: ContraBand implants

INTERVENTIONS:
Device: ContraBand implants — Percutaneous implantation of the ContraBand devices by right heart catheterization

SUMMARY:
ContraBand™ is a transcatheter constriction device which is implanted in the left and right branch pulmonary arteries. The effect is achieved by causing a local reduction in the internal diameters of the branch PAs, resulting in a lower distal systolic pulmonary artery pressure (PAP) as well as an attenuation in the rise of the mean pulmonary capillary wedge pressure (PCWP) along with a higher pulmonary arterial compliance (PAC) distal to the constriction during exercise. Lower PCWP reflects the reduced left ventricular end diastolic pressure (LVEDP), contributing to enhanced ventricular filling and improved cardiac output. This hemodynamic change is anticipated to translate into enhanced physical capacity and a potentially more favorable prognosis for heart failure subjects. This study is an early feasibility, multi center, prospective, interventional, open-label, single-arm study.

ELIGIBILITY:
Main Inclusion Criteria:

* Age is 18 - 85 years old
* Chronic heart failure (> 3 months)
* Symptomatic left heart failure Stage C (NYHA Class III-IVa) or Class II with documented prior history of Class III-IVa heart failure.
* LVEF 20 - 40%
* Receiving optimally tolerated GDMT for at least 3 (three) months as referred in the 2021 ESC Guidelines for the optimal recommended pharmacological treatment indicated in patients with (NYHA class II-IV) heart failure with reduced ejection fraction (LVEF< 40%).
* If indicated according to the 2021 ESC Guidelines: Subject has an implantable cardioverter-defibrillator (ICD) for at least 1 month prior to screening. or subject is on cardiac resynchronization therapy (CRT)/pacemaker for at least 3 months prior to screening.
* Able to complete six-minute walk test (6MWT) with distance between 100 meters and 400 meters.

Main Exclusion Criteria:

* Serum NT-proBNP <300 pg/mL
* Significant RV dysfunction with TAPSE < 15 mm
* Moderate to severe pulmonary hypertension (Pulmonary vascular resistance PVR ≥ 4.0 WU and PAPi < 1.0 by RHC)
* Anatomical pathology or constraints preventing appropriate access/implant of ContraBand™
* Restrictive Cardiomyopathy or myocarditis
* Any severe valve disease (Grade 3-4) and/or tricuspid regurgitation ≥ 2+ (in a scale of 5)
* Hemodynamic instability: Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or mechanical hemodynamic support
* Active bacterial endocarditis or previous history of SBE (Subacute bacterial endocarditis)
* Any planned cardiac surgery or interventions within the next six (6) months
* Need for coronary artery revascularization
* Myocardial infarction or any percutaneous cardiovascular intervention within 1 month
* Cardiovascular surgery, or carotid surgery within 3 months
* Acute kidney insufficiency and/or end stage renal disease requiring chronic dialysis (eGFR < 30)
* Leukopenia (WBC < 4000 cells/μL), anemia (Hgb < 9 g/dL), thrombocytopenia (platelets < 150,000 cells/μL) or any known blood clotting disorder
* History of systemic or pulmonary thromboembolism within 12 months prior to Baseline visit; incidental small peripheral pulmonary emboli deemed clinically insignificant by the investigator are not considered exclusionary
* Previous history of cardiogenic shock (unrelated to myocardial infraction)
* Stroke, transient ischemic attack (TIA) or deep vein thrombosis (DVT) within 6 months of screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-related or procedure-related major adverse events (MAEs) | 30 days
  MAE is a composite of death; myocardial infarction; emergent conversion to surgery; stroke; major cardiac structure complication; major vascular complication; embolization and heart failure- related hospitalization.

SECONDARY OUTCOMES:
Procedural success | Implantation procedure
  Ability to successfully deliver devices to the Pulmonary Arteries

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (3):
  - Clinical Site, Aalst
  - Clinical Site, Antwerp
  - Clinical Site, Genk
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia
- Clinical Site, Lübeck, Germany
- Israel (3):
  - Clinical Site, Nahariya
  - Clinical Site, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Lithuania (2):
  - Clinical Site, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (2):
  - Clinical Site, Krakow
  - Clinical Site, Lublin

IPD SHARING:
Plan to Share IPD: No